CLINICAL TRIAL: NCT00334724
Title: Home Blood Pressure-guided Antihypertensive Intervention for Elderly (HBP-GUIDE) Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Patients were not appropriately enrolled
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Collaborators: Kyoto Prefectural University of Medicine (Other)
Responsible Party: Hiroaki Matsubara, Kyoto Prefectural University of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-136
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Disease; Vascular Disease; Hypertension
Keywords: Cardiovascular disease; Vascular disease; Hypertension; Home blood pressure measurement
MeSH Terms: conditions — Cardiovascular Diseases; Vascular Diseases; Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Home blood pressure group
  Interventions: Procedure: Home blood pressure measurement
- 2 (Active Comparator): Office blood pressure group
  Interventions: Procedure: Office blood pressure measurement

INTERVENTIONS:
Procedure: Home blood pressure measurement — Blood pressure controlled based on home blood pressure measurement
  Arms: 1
Procedure: Office blood pressure measurement — Blood pressure controlled based on office blood pressure measurement
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether blood pressure control by home blood pressure monitoring exerts beneficial cardioprotective effects rather than by clinic blood pressure monitoring in elderly patients.

DETAILED DESCRIPTION:
Home blood pressure (BP) measurement has been reported to be closely correlated with target organ damage and appears to be a prognostic indicator with respect to cardiovascular mortality and cardiovascular events. However, whether BP control by home BP monitoring exerts cardioprotective effects rather than by clinic BP monitoring in elderly patients remains unknown. In this study, a total of 500 elderly patients diagnosed with essential hypertension will be randomly divided into 2 groups; target BP level, home SBP <135 mmHg and home DBP <85 mmHg (home BP control group), clinic SBP <140 mmHg and clinic DBP <90 mmHg (clinic BP control group). Olmesartan at doses of 20 mg/day will be administered and increased up to 40 mg, if antihypertensive effect is inadequate. Study visits will be made bimonthly for at least 1 year. The antihypertensive and cardioprotective effects including systemic levels of C-reactive protein and inflammatory cytokines, and arterial stiffness will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged over 65 years and less than 80 years
* Patients with a stable seated systolic blood pressure of ≥ 140 mmHg or diastolic blood pressure of ≥ 90 mmHg at two visits within 8 weeks
* Patients with a stable seated systolic blood pressure of ≥ 135 mmHg or diastolic blood pressure of ≥ 85 mmHg at home (home blood pressure is measured every morning within 1 h of waking, and defined as the mean of 3 days measurement within 8 weeks)

Exclusion Criteria:

* Patients with secondary hypertension or malignant hypertension
* Patients with a stable seated systolic pressure of ≥ 180 mmHg or diastolic pressure of ≥ 110 mmHg
* Patients with renal dysfunction with a serum creatinine level of ≥ 2 mg/dl
* Patients with liver dysfunction
* Patients with a history of hypersensitivity to angiotensin II receptor blockade
* Patients with a history of myocardial infarction within 6 months prior to enrolment in the study
* Patients who underwent coronary arterioplasty within 6 months prior to enrolment in the study or patients who will undergo coronary arterioplasty within 6 months after entry
* Patients with heart failure
* Patients with a history of cerebrovascular disorder
* Other patients who are judged to be inappropriate for the study by the investigator

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Home blood pressure | one year
Office blood pressure | one year

SECONDARY OUTCOMES:
high sensitive C-reactive protein | one year
Interleukin-6 | one year
urine microalbumin | one year
Plasminogen activator inhibitor activity | one year
B-type natriuretic peptide | one year
Pulse wave velocity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Matsubara, MD, PhD, Principal Investigator — Professor of Medicine, Department of Cardiovascular Medicine, Kyoto Prefectural University of Medicine
Locations (1):
- Division of Internal Medicine, Kyoto Prefectural University of Medicine, Kyoto, Kyoto, Japan